CLINICAL TRIAL: NCT03377270
Title: Clinical Impact of Respiratory-Swallow Training on Refractory Dysphagia in OP HNC
Brief Title: Clinical Impact of Respiratory-Swallow Training on Refractory Dysphagia in Oropharyngeal Head and Neck Cancer
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: VA Office of Research and Development (U.S. Federal Agency)
Collaborators: Edward Hines Jr. VA Hospital (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: F2352-R
Record Dates: First submitted 2017-12-08; First posted 2017-12-19 (Actual); Results first posted 2025-05-06 (Actual); Last update posted 2025-05-06 (Actual); Status verified 2025-04

CONDITIONS: Head and Neck Cancer; Dysphagia
Keywords: Oropharyngeal Head and Neck Cancer; dysphagia; Respiratory Swallow Training
MeSH Terms: conditions — Head and Neck Neoplasms; Deglutition Disorders

STUDY DESIGN:
Intervention Model Description: Randomized-controlled trial with 2 arms (intervention and control)
Who Masked: Outcomes Assessor
Masking Description: outcomes assessor (those completed the swallow studies, those scoring)
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Arm 1. Immediate Respiratory-Swallow Training (Experimental): Description: Participants receive Respiratory-Swallow Training (RST) immediately after baseline evaluation. RST retrains swallowing initiation to occur during exhalation at mid-to-low lung volumes.
  Intervention Schedule: Begins within 1 week of baseline evaluation and continues for 4 weeks (two 1-hour sessions per week).
  Post-RST Assessment: Conducted within 1-week post-intervention and at 1-, 3-, and 6-months to assess efficacy and durability.
  Interventions: Behavioral: Respiratory Swallow Training
- Arm 2. Delayed Respiratory-Swallow Training (Other): Description: Participants receive no active intervention for the first 4 weeks post-baseline, then begin Respiratory-Swallow Training (RST) using the same protocol as Arm 1.
  Intervention Schedule: Begins 4 weeks after baseline evaluation and continues for 4 weeks (two 1-hour sessions per week).
  Post-RST Assessment: Conducted within 1-week post-intervention and at 1-, 3-, and 6-months to assess efficacy and durability.
  Interventions: Behavioral: Respiratory Swallow Training

INTERVENTIONS:
Behavioral: Respiratory Swallow Training — Training in the Optimal Respiratory Swallow Pattern and Lung Volume at Swallow Initiation

SUMMARY:
Veterans following treatment of head and neck cancer can be left with lasting swallowing impairment that may require diet alterations, need for feeding tubes, and risk of pneumonia. The investigators' previous trial tested a new swallowing treatment approach to target respiratory-swallow coordination. The results revealed improvements in respiratory-swallow coordination and swallowing function. The goal of this study is to determine the impact and durability of respiratory-swallow training (RST) on clinical outcomes necessary for eating, drinking, health, and quality-of-life in Veterans with swallowing impairment following treatment for head and neck cancer. A total of 50 participants will be recruited with a goal of 40 randomly assigned to immediate RST or delayed RST.

DETAILED DESCRIPTION:
Head and neck cancer (HNC) is a significant health issue in Veterans. In fact, Veterans have up to a two-fold increase in the incidence of HNC when compared to the general population. Further, they often suffer profound functional deficits associated with surgical ablation and toxicity from medical treatments used to cure or control local disease. Dysphagia (swallowing impairment) is common after such treatments, and has life-altering consequences [on health, quality-of-life, the ability to eat and drink normally, cost, and burden of care]. Despite important advancements in medical and surgical treatments that prolong survival, many Veterans with HNC, are faced with chronic, intractable dysphagia resulting in persistent drastic alterations in diet, the need for feeding tubes, and increased risk for aspiration pneumonia - a life threatening infection. The investigators must devote research and clinical efforts to mitigate these devastating impairments because the investigators' current rehabilitative intervention options are severely limited. As such, and in keeping with the VHA's Blueprint for Excellence Transformative Actions, the need for the development of effective swallowing interventions that show potential for rapid translation to clinical practice is imperative.

Coordination of respiration and swallowing is an essential element of airway protection during swallowing and facilitates many critical aspects of swallowing physiology. This key, coordinative event is significantly disrupted in patients with dysphagia following medical and surgical treatments for HNC. The investigators' previous trial in patients with severe and resistant dysphagia after cancer treatment and traditional swallowing therapy showed that targeting and recalibrating respiratory-swallow phase patterning directly through an innovative respiratory-swallow training (RST) method significantly improved aspects of swallowing physiology crucial for airway protection and clearance of ingested materials through the pharynx. These exciting new results led us to consider an expanded study with refined methods and a home practice (HP) component that will extend beyond physiologic efficacy and include more rigorous assessments of the clinical impact of RST. As with the investigators' preliminary trial, the investigators' prediction is that these innovative intervention methods will not only improve swallowing physiology and quality-of-life, but will also result in significant functional improvements in every day eating and drinking in Veterans with chronic, severe dysphagia that has been otherwise refractory to traditional swallowing intervention(s). The benefit of RST training is that it is a simple, straightforward method for patients to easily learn, and, when combined with the HP program, it is designed to facilitate patient compliance and maintenance of intervention effects. The investigators are also using commercially available and simple to use recording and analysis hardware and software that can easily be expanded to mobile technology for more widespread application to the many thousands of patients with dysphagia consequent to HNC.

A total of 50 participants will be recruited with the goal of 40 participants enrolled. Participants will be randomly assigned 1:1 to either immediate RST (intervention arm) or delayed RST (control arm). The participants in the control arm will have no active treatment for 4 weeks and will then participate in RST as a cross-over design. Data obtained will be used to evaluate clinical efficacy and durability The primary efficacy endpoint is physiologic function metrics of the oropharyngeal swallow, and the secondary endpoints are airway invasion and patient reported outcomes. We will use reproducible, reliable, and validated metrics that include the Modified Barium Swallow Impairment Profile and Penetration-Aspiration Scale to distinguish the mechanistic effects of RST.

The goal of this current study is to extend the investigator's preliminary trial that yielded compelling physiologic changes with potential to improve the impact and durability of RST on clinical outcomes essential for eating, drinking, health, and quality-of-life. The investigators' overarching goal is to provide two parallel tracks of knowledge generation: 1) provide immediate clinical translation of experimental findings to improve the lives of Veterans, and 2) drive model generation on fundamental mechanisms of motor coordination. Basic knowledge will drive clinical application and vice-a-versa. As such, this is an ideal experimental and clinical context that will fuel knowledge generation in this highly significant area of science and clinical practice.

ELIGIBILITY:
Inclusion Criteria:

* Veteran and non Veterans
* have undergone treatment for a primary diagnosis of head and neck cancer (oral cavity, oropharyngeal, and hypopharyngeal)
* are 21 years of age
* 6 months post head and neck cancer treatment
* 6 months post-traditional swallowing treatment with continued dysphagia
* English speaking
* pass a cognitive screening (score 26 on the Montreal Cognitive Assessment (MoCA)
* do not present with severe chronic obstructive pulmonary disease (COPD) based on pulmonary function testing (PFT)
* drink less than 2 alcoholic beverages per day

Exclusion Criteria:

* if they have known allergy or dietary restriction for contrast materials or liquids used during the MBSS or training
* currently drinking greater than two drinks per day
* severe COPD
* are unable to swallow one liquid consistency without the use of a compensatory strategy or swallow maneuver without aspiration
* history of aspiration pneumonia within the past 12 months

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 49 (Actual)
Dates: Start 2018-10-01 (Actual); Primary Completion 2023-12-31 (Actual); Study Completion 2023-12-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Bonnie J. Martin-Harris, PhD, Principal Investigator — Edward Hines Jr. VA Hospital, Hines, IL
Locations (2):
- United States (2):
  - Northwestern University, Chicago, Illinois
  - Edward Hines Jr. VA Hospital, Hines, IL, Hines, Illinois

IPD SHARING:
Plan to Share IPD: No
All participants' data will be de-identified and aggregated for analysis

RESULTS

PARTICIPANT FLOW:
Period: Intervention RST
Arm/Group | Arm 1. Immediate Respiratory-Swallow Training | Arm 2. Delayed Respiratory-Swallow Training
Started | 28 | 21
Completed | 26 | 15
Not Completed | 2 | 6
Period: Follow Up
Arm/Group | Arm 1. Immediate Respiratory-Swallow Training | Arm 2. Delayed Respiratory-Swallow Training
Started | 26 | 15
Completed | 25 | 13
Not Completed | 1 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Arm 1. Immediate Respiratory-Swallow Training | Arm 2. Delayed Respiratory-Swallow Training | Total
Number analyzed (Participants) | 28 | 21 | 49
Age, Continuous [Mean (Full Range); unit: years] | 65 [48 to 79] | 66 [48 to 77] | 65 [48 to 79]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 4 | 6
  Male | 26 | 17 | 43
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 0 | 1
  Not Hispanic or Latino | 27 | 21 | 48
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 2 | 2
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 3 | 4 | 7
  White | 24 | 15 | 39
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 1 | 0 | 1

OUTCOME MEASURES:

1. Primary Outcome: Modified Barium Swallow Impairment Profile (MBSImP) Pharyngeal Total (PT) Score
Description: The MBSImP is a standardized outcome measure that evaluates swallowing physiology using 17 distinct component scores across the oral (components 1-6), pharyngeal (components 7-16), and esophageal (component 17) domains. Each component is rated on an ordinal scale based on specific physiologic impairments. Scores range from a minimum of 0 (no impairment) to a maximum of 2, 3, or 4, depending on the component. Higher scores indicate greater swallowing dysfunction, reflecting worse outcomes. For this analysis, the pharyngeal total (PT) score was used as a primary outcome measure. The PT score provides a comprehensive measure of overall pharyngeal function and is a sum of components 7 through 16. The PT Score ranges from 0 to 32, with higher scores indicating greater severity of impairment in pharyngeal swallowing function. A score of 0 represents no impairment, while a score of 32 represents the most severe impairment.
Time Frame: Baseline, 30 days, 60 days, 120 days, 240 days
Population: Of the 49 subjects who entered the intervention phase, 40 were included in the final analysis. Nine participants withdrew.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Arm 1. Immediate Respiratory-Swallow Training | Arm 2. Delayed Respiratory-Swallow Training
Number analyzed (Participants) | 25 | 15
score on a scale
  Baseline | 11.00 (4.70) | 12.33 (4.62)
  30 days | 9.84 (4.01) | 10.73 (4.77)
  60 days | 10.17 (4.66) | 11.00 (5.08)
  120 days | 10.45 (3.66) | 10.17 (5.39)
  240 days | 12.23 (3.98) | 11.50 (5.37)

2. Secondary Outcome: Maximum Penetration Aspiration Scale (PAS) Score
Description: Measures the presence, depth, and reaction to penetration and aspiration during swallowing as observed through videofluoroscopy. The PAS is scored on an 8-point ordinal scale, with values ranging from 1 (no airway entry) to 8 (silent aspiration, with material passing below the vocal folds and no response). Higher scores indicate greater severity of airway compromise, reflecting worse outcomes in terms of swallowing safety.
Time Frame: Baseline, 30 days, 60 days, 120 days, 240 days
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Arm 1. Immediate Respiratory-Swallow Training | Arm 2. Delayed Respiratory-Swallow Training
Number analyzed (Participants) | 25 | 15
score on a scale
  Baseline | 4.16 (2.44) | 4.73 (2.58)
  30 days | 3.68 (2.43) | 3.60 (1.99)
  60 days | 4.17 (2.62) | 3.92 (2.33)
  120 days | 3.77 (2.58) | 4.67 (2.19)
  240 days | 4.55 (2.61) | 4.42 (2.31)

3. Secondary Outcome: MD Anderson Dysphagia Inventory (MDADI) Composite Score
Description: A patient-reported outcome measure designed to assess the impact of dysphagia on quality of life in individuals with head and neck cancer. The MDADI includes 20 items scored across three subscales: Emotional, Functional, and Physical. Each item is rated on a 5-point Likert scale (1 = strongly agree to 5 = strongly disagree), with lower scores indicating worse quality of life related to dysphagia. The Composite Score is calculated by summing the scores from the Emotional, Functional, and Physical subscales. A score of 20 indicates the worst possible quality of life related to dysphagia, while a score of 100 indicates the best possible quality of life.
Time Frame: Baseline, 30 days, 60 days, 120 days, 240 days
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Arm 1. Immediate Respiratory-Swallow Training | Arm 2. Delayed Respiratory-Swallow Training
Number analyzed (Participants) | 25 | 15
score on a scale
  Baseline | 63.33 (16.83) | 59.40 (12.67)
  30 days | 64.17 (16.81) | 64.62 (18.76)
  60 days | 66.63 (19.25) | 67.45 (19.08)
  120 days | 67.03 (20.93) | 70.53 (17.22)
  240 days | 68.74 (17.49) | 71.49 (18.81)

4. Secondary Outcome: Functional Oral Intake Scale (FOIS) Score
Description: Assesses the level of oral intake in individuals with dysphagia. The FOIS is scored on a 7-point ordinal scale, ranging from 1 (nothing by mouth) to 7 (full oral intake with no restrictions). Higher scores indicate better functional oral intake and less dependence on alternative feeding methods.
Time Frame: Baseline, 30 days, 60 days, 120 days, 240 days
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Arm 1. Immediate Respiratory-Swallow Training | Arm 2. Delayed Respiratory-Swallow Training
Number analyzed (Participants) | 25 | 15
score on a scale
  Baseline | 5.56 (1.19) | 5.43 (0.94)
  30 days | 5.56 (1.16) | 5.67 (1.23)
  60 days | 5.64 (0.95) | 5.64 (1.12)
  120 days | 5.68 (0.95) | 5.83 (1.11)
  240 days | 5.86 (1.31) | 6.09 (0.83)

5. Secondary Outcome: Performance Status Scale for Head and Neck Cancer (PSS-HN) Subscales Scores
Description: Evaluates the functional impact of head and neck cancer on patients' ability to eat and communicate. The PSS-HN includes three subscales: Normalcy of Diet, Understandability of Speech, and Eating in Public, each scored on a 0-100 scale, with higher scores indicating better performance and less functional impairment.
Time Frame: Baseline, 30 days, 60 days, 120 days, 240 days
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Arm 1. Immediate Respiratory-Swallow Training | Arm 2. Delayed Respiratory-Swallow Training
Number analyzed (Participants) | 25 | 15
score on a scale
  Baseline PSS-HN Diet | 59.60 (21.31) | 60.77 (21.39)
  30 days PSS-HN Diet | 60.50 (20.64) | 67.27 (24.53)
  60 days PSS-HN Diet | 60.00 (20.29) | 61.11 (22.05)
  120 days PSS-HN Diet | 63.75 (20.29) | 68.00 (23.00)
  240 days PSS-HN Diet | 69.52 (22.02) | 78.00 (22.51)
  Baseline PSS-HN Public | 73.96 (32.54) | 85.42 (22.51)
  30 days PSS-HN Public | 73.75 (31.91) | 81.82 (27.59)
  60 days PSS-HN Public | 77.94 (23.19) | 72.22 (34.11)
  120 days PSS-HN Public | 76.56 (28.09) | 82.50 (31.29)
  240 days PSS-HN Public | 76.19 (29.02) | 90.91 (20.23)
  Baseline PSS-HN Speech | 92.71 (13.75) | 85.42 (12.87)
  30 days PSS-HN Speech | 90.00 (17.01) | 90.91 (12.61)
  60 days PSS-HN Speech | 89.71 (17.81) | 93.75 (11.57)
  120 days PSS-HN Speech | 92.19 (15.05) | 85.00 (21.08)
  240 days PSS-HN Speech | 92.86 (14.02) | 88.64 (13.06)

ADVERSE EVENTS:
Time Frame: 240 days
Description: This two-arm RCT was designed to assess the timing of Respiratory-Swallow Training (RST) on swallowing outcomes. All participants received RST; the only difference was when it began. Arm 1 received RST immediately; Arm 2 after a 4-week delay reflecting standard care in patients with chronic dysphagia post-HNC. Adverse events are attributed by assigned arm. Adding a third "no-treatment" arm would inaccurately suggest a subgroup of participants who received no intervention at all.
Arm/Group | Arm 1. Immediate Respiratory-Swallow Training | Arm 2. Delayed Respiratory-Swallow Training
All-Cause Mortality (participants affected / at risk) | 0/28 | 0/21
Serious Adverse Events (participants affected / at risk) | 0/28 | 1/21
Other Adverse Events (participants affected / at risk) | 0/28 | 0/21
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Arm 1. Immediate Respiratory-Swallow Training (N=28) | Arm 2. Delayed Respiratory-Swallow Training (N=21)
Cerebrovascular Accident (CVA) (Nervous system disorders) | 0 (0) | 1 (1) — Unrelated to the participant's participation in the research.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2023-01-24): https://cdn.clinicaltrials.gov/large-docs/70/NCT03377270/Prot_SAP_000.pdf
  • Informed Consent Form (2023-01-05): https://cdn.clinicaltrials.gov/large-docs/70/NCT03377270/ICF_001.pdf